CLINICAL TRIAL: NCT02423616
Title: Correlation Between Maximal Inspiratory Pressure and Hand Grip Force in Healthy Individuals
Brief Title: Correlation Between Maximal Inspiratory Pressure and Hand Grip Force
Acronym: CBMIPHGFHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Efstathiou Ioannis, Efstathiou Ioannis .P.T, Attikon Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 3-13/11-2-16
Record Dates: First submitted 2015-04-04; First posted 2015-04-22 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: MIP; Hand Grip; Correlation; Inspiratory Pressure; Hand Grip Force

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy individuals (Experimental): Study population was consisted by healthy volunteers from hospital staff of physical therapy department, Intensive Care Unit, and cleaning service. All subjects were men and women aged between 20 and 65 years old, who never had major problems with the respiratory system or with the hand flexors.
  Interventions: Other: Healthy individuals

INTERVENTIONS:
Other: Healthy individuals — INSPIRATORY PRESSURE AND HAND GRIP FORCE CORRELATION

SUMMARY:
This study aimed to examine the possible relationship between hand grip strength (HGS) and maximum inspiratory pressure (MIP) in healthy individuals.

DETAILED DESCRIPTION:
This study aimed to examine the possible relationship between hand grip strength (HGS) and maximum inspiratory pressure (MIP) in healthy individuals. All individuals underwent assessment of inspiratory muscle strength by maximum inspiratory pressure, and evaluation of hand grip strength. MIP was measured using a U-type water manometer calibrated in centimetre of water (cmH2O), while the HGS was measured with hydraulic hand dynamometer calibrated in Kg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* age <20 years old,
* pregnancy,
* official diagnosis with lung disease such as Chronic obstructive pulmonary disease (COPD),
* body mass index (BMI) > 40,
* known pre-existing causes of neuromuscular weakness,
* median entrapment neuropathy such as carpal tunnel syndrome

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
CORRELATION BETWEEN MAXIMAL INSPIRATORY PRESSURE AND HAND GRIP FORCE | one month
  MIP was measured using a U-type water manometer calibrated in cmH2O, while the HGS was measured with hydraulic hand dynamometer calibrated in Kg.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Armaganidis, M.D, Study Chair — Univercity of Athens; Eirine Maurou, MD, Study Director — Attikon Hospital; Konstantinos Grigoriadis, PT, MSc, Study Director — Attikon Hospital; Ioannis Efstathiou, PT, Principal Investigator — Attikon Hospital; Eirini Maurou, MD, Study Director — Attikon Hospital

REFERENCES:
- [Background] Larson JL, Covey MK, Vitalo CA, Alex CG, Patel M, Kim MJ. Maximal inspiratory pressure. Learning effect and test-retest reliability in patients with chronic obstructive pulmonary disease. Chest. 1993 Aug;104(2):448-53. doi: 10.1378/chest.104.2.448. PMID 8339633
- [Derived] Efstathiou ID, Mavrou IP, Grigoriadis KE. Correlation Between Maximum Inspiratory Pressure and Hand-Grip Force in Healthy Young and Middle-Age Individuals. Respir Care. 2016 Jul;61(7):925-9. doi: 10.4187/respcare.04319. Epub 2016 Apr 19. PMID 27094394